CLINICAL TRIAL: NCT01709045
Title: The Assessment of the Plaque at RISK by Non-invasive (Molecular) Imaging and Modelling (ParisK): Correlation of Imaging Techniques With Histology
Brief Title: ParisK: Correlation of Imaging Techniques With Histology
Acronym: ParisK
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Center for Translational Molecular Medicine (Other); Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 10-2-048
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Plaque, Atherosclerotic
Keywords: Endarterectomy, Carotid; Carotid Arteries
MeSH Terms: conditions — Stroke; Plaque, Atherosclerotic | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Carotid plaque removed during carotid endarterectomy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients scheduled for CEA: All patients who are scheduled for carotid endarterectomy (CEA)
  Interventions: Other: Magnetic Resonance Imaging (MRI); Radiation: Dual-Energy Computed Tomography (DECT); Other: Ultrasound; Other: Transcranial doppler

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — Multi-sequence MR protocol
  Other Names: 3.0 T Philips Achieva
Radiation: Dual-Energy Computed Tomography (DECT)
  Other Names: Siemens Flash
Other: Ultrasound
  Other Names: Philips IU22
Other: Transcranial doppler
  Other Names: Hemodynamics AG

SUMMARY:
The possibility to identify the risk of rupture of a carotid plaque will have tremendous impact in clinical decision making. A vulnerable plaque is considered to have a large lipid rich necrotic core (LRNC), a thin fibrous cap, the presence of inflammatory cells, intraplaque haemorrhage and/or neovascularisation (vasa vasorum). The investigators aim to validate imaging of plaque vulnerability with histology. Previous studies have evaluated the use of imaging to assess carotid plaque vulnerability, mostly showing a good correlation between imaging and histology and/or clinical characteristics. However, they have focused on single modalities, (magnetic resonance imaging [MRI], multidetector-row computed tomography (MDCT), ultrasonography (US) or transcranial Doppler (TCD), and have used relatively small cohorts

The primary goal of this study is to investigate whether there is a correlation between neovascularisation in the carotid atherosclerotic plaque as observed with 3.0 Tesla dynamic contrast-enhanced MRI and histology. Moreover, the investigators aim to investigate the correlation between the volume of the LRNC as determined by dual-energy CT and histology.

Secondly, the investigators will investigate the correlation between the volume of the LRNC, the fibrous cap status and the volume of the calcifications determined by MRI versus histology, the correlation between number of microembolisms and fibrous cap status and the correlation between the deformation pattern seen with ultrasound and the volume of the LRNC.

The imaging parameters showing good correlation with plaque vulnerability characteristics can be used for further analysis in assessing the vulnerable plaque

ELIGIBILITY:
Inclusion Criteria:

* Patients with a carotid artery stenosis, who are scheduled for carotid endarterectomy
* Age 18 years or older (no maximum age)
* Informed consent by signing informed consent form regarding this study
* Inclusion criteria for carotid endarterectomy

  1. Symptomatic carotid artery stenosis 70-99% within 3 months of neurological symptoms
  2. Symptomatic carotid artery stenosis 50-99% in man within 2 weeks of neurological symptoms
  3. Asymptomatic carotid artery stenosis 70-99% with contralateral occlusion

Exclusion Criteria:

* Severe co-morbidity, dementia or pregnancy
* Standard contra-indications for MRI (ferromagnetic implants like pacemakers or other electronic implants, metallic eye fragments, vascular clips, claustrophobia, etc.)
* Patients who have a documented allergy to MRI or CT contrast media
* Patients with a renal clearance <30 ml/min are not eligible to undergo contrast-enhanced MRI
* Patients with a renal clearance <60 ml/min are not eligible to undergo CT
* Surgery planned within 4 days of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a carotid artery stenosis, who are scheduled for carotid endarterectomy, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Ktrans on dynamic contrast-enhanced (DCE)-MRI | 1 day
  The correlation between neovascularisation in carotid atherosclerotic plaque as assessed by dynamic 3.0 Tesla MRI and microvasculature as assessed by histology.
Lipid-rich necrotic core on dual-energy CT | 1 day
  The correlation between the size of lipid-rich-necrotic-core in dual-energy CT and histology.

SECONDARY OUTCOMES:
deformation pattern on ultrasound | 1 day
  The correlation between deformation pattern at echo and plaque composition (volume of LRNC) at histology.
number of recorded micro embolic signals (MES) | 1 day
  The relation between number of recorded MES and fibrous cap status at histology.
Volume of LRNC and calcifications and fibrous cap status on MRI | 1 day
  The correlation between volume of LRNC, fibrous cap status and volume of calcifications in carotid atherosclerotic plaques visualised by MRI and the same features as determined at histology.

CONTACTS AND LOCATIONS:
Overall Officials: Eline Kooi, PhD, Study Chair — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Aizaz M, Bierens J, Gijbels MJJ, Schreuder THCML, van Orshoven NP, Daemen JHC, Mess WH, Flohr T, van Oostenbrugge RJ, Postma AA, Kooi ME. Differentiation of Atherosclerotic Carotid Plaque Components With Dual-Energy Computed Tomography. Invest Radiol. 2025 Aug 1;60(8):508-516. doi: 10.1097/RLI.0000000000001153. Epub 2025 Jan 22. PMID 39836610
- [Derived] Crombag GAJC, Schreuder FHBM, van Hoof RHM, Truijman MTB, Wijnen NJA, Voo SA, Nelemans PJ, Heeneman S, Nederkoorn PJ, Daemen JH, Daemen MJAP, Mess WH, Wildberger JE, van Oostenbrugge RJ, Kooi ME. Microvasculature and intraplaque hemorrhage in atherosclerotic carotid lesions: a cardiovascular magnetic resonance imaging study. J Cardiovasc Magn Reson. 2019 Mar 4;21(1):15. doi: 10.1186/s12968-019-0524-9. PMID 30832656
- [Derived] Truijman MT, de Rotte AA, Aaslid R, van Dijk AC, Steinbuch J, Liem MI, Schreuder FH, van der Steen AF, Daemen MJ, van Oostenbrugge RJ, Wildberger JE, Nederkoorn PJ, Hendrikse J, van der Lugt A, Kooi ME, Mess WH; Plaque at RISK Study. Intraplaque hemorrhage, fibrous cap status, and microembolic signals in symptomatic patients with mild to moderate carotid artery stenosis: the Plaque at RISK study. Stroke. 2014 Nov;45(11):3423-6. doi: 10.1161/STROKEAHA.114.006800. Epub 2014 Sep 25. PMID 25256179